CLINICAL TRIAL: NCT00550277
Title: A Phase II Study of LBH589 in the Treatment of Patients With Refractory Clear Cell Renal Carcinoma
Brief Title: LBH589 Treatment for Refractory Clear Cell Renal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 49
Record Dates: First submitted 2007-10-26; First posted 2007-10-29 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Refractory; LBH589
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): LBH589 will be administered orally at a dose of 45 mg (1 - 5 mg capsule and 2 - 20 mg capsules) on Monday and Thursday of each week (twice weekly). To enable patients to undergo cardiac monitoring, all patients must begin treatment on a Monday, and continue Monday/Thursday dosing during subsequent treatment cycles. Patients with objective response or stable disease after re-evaluation at week 8 will continue LBH589 at the same dose until disease progression, unacceptable toxicity and/or at the discretion of the investigator.
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589 — LBHLBH589 will be administered orally at a dose of 45 mg (1 - 5 mg capsule and 2 - 20 mg capsules) on Monday and Thursday of each week (twice weekly). To enable patients to undergo cardiac monitoring (Section 3.5.2), all patients must begin treatment on a Monday, and continue Monday/Thursday dosing during subsequent treatment cycles.
  Other Names: Panobinostat

SUMMARY:
Inhibition of histone deacetylase (HDAC) provides a novel approach for cancer treatment. LBH589, an oral HDAC inhibitor, has been well tolerated in phase I trials and has shown activity against several types of cancer. In this nonrandomized phase II trial, we are investigating the activity of LBH589 in the treatment of patients with refractory clear cell renal carcinoma.

DETAILED DESCRIPTION:
Inhibition of histone deacetylase (HDAC) provides a potential target for cancer treatment. Histones are components of the core proteins of nucleosomes, and acetylation and deacetylation of these proteins play a role in the regulation of gene expression. HDAC activity is known to be increased in many types of malignant cells; HDAC inhibitors have been shown to induce differentiation, cell cycle arrest, and apoptosis in cultured tumor cells. Since this tumor-associated mechanism is common to many types of cancer, HDAC may have a broad role in cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented metastatic or locally unresectable clear cell renal carcinoma. In patients with mixed histologies, the clear cell component must comprise > 75% of the cancer.
* Documented disease progression or intolerance while receiving treatment with: a) sunitinib, sorafenib, or both, and b) temsirolimus.
* Maximum of 4 prior systemic regimens allowed and may include other targeted agents, immunotherapy and chemotherapy.
* Measurable disease by RECIST criteria.
* ECOG PS 0 or 1.
* Laboratory values as follows: ANC >= 1500/μL, Hgb >= 9 g/dL, Platelets >= 100,000/uL, AST/SGOT and ALT/SGPT <= 2.5 x ULN or <= 5.0 x ULN in patients with liver metastases, Creatinine <= 2.0 mg/dL Or Calculated Creatinine Clearance >= 50 ml/min, Albumin >= 3 g/dL, Potassium >= lower limit normal (LLN),Phosphorous >= LLN, Calcium >= LLN, Magnesium > LLN
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment.
* Life expectancy > 12 weeks.
* Accessible for treatment and follow-up.
* All patients must be able to understand the nature of the study and give written informed consent prior to study entry.

Exclusion Criteria:

* Age < 18 years of age.
* Prior treatment with an HDAC inhibitor.
* Impaired cardiac function
* Ongoing therapy with antiarrhythmics or other medications associated with QTc prolongation.
* Uncorrected hypokalemia or hypomagnesemia.
* Uncontrolled hypertension or cardiac arrhythmias.
* Active parenchymal brain metastases. Patients who have had brain metastases resected, or have received radiation therapy ending > 8 weeks prior to study entry are eligible if they meet all of the following criteria: 1) residual neurologic symptoms < grade 1, 2) no dexamethasone requirement, 3) follow-up MRI shows regression of lesions after treatment, with no new lesions appearing.
* Active meningeal metastases.
* Known diagnosis of human immunodeficiency virus (HIV) infection.
* Unresolved diarrhea > CTCAE grade 1.
* Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors.
* Chemotherapy, investigational drug therapy, major surgery < 4 weeks prior to starting study drug or patients that have not recovered from side effects of previous therapy.
* Patient is < 5 years free of another primary malignancy except if the other primary malignancy is not currently clinically significant or requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Concomitant use of any anti-cancer therapy or radiation therapy.
* Pregnant or breast feeding or female of reproductive potential not using 2 effective methods of birth control.
* Male patients whose sexual partners are women of childbearing potential not using effective birth control.
* Patients with gastrointestinal (GI) tract disease, causing the inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease.
* Other concurrent severe, uncontrolled infection or intercurrent illness
* Abnormal thyroid function (TSH or free T4) detected at screening. Patients with known hypothyroidism who are stable on thyroid replacement are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (10):
- United States (10):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Methodist Cancer Center, Omaha, Nebraska
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia

REFERENCES:
- [Background] Hainsworth JD, Infante JR, Spigel DR, Arrowsmith ER, Boccia RV, Burris HA. A phase II trial of panobinostat, a histone deacetylase inhibitor, in the treatment of patients with refractory metastatic renal cell carcinoma. Cancer Invest. 2011 Aug;29(7):451-5. doi: 10.3109/07357907.2011.590568. Epub 2011 Jun 22. PMID 21696296

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 20
Completed | 11
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the interval from the date of first treatment with panobinostat until the date that disease progression or death occurred. Progressive disease (PD): 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 20
months | 1.7 [1.2 to 2.6]

2. Secondary Outcome: Number of Participants Experiencing ≥Grade 2 Adverse Events
Description: An adverse event (AE) is the development of an undesirable medical condition, or the deterioration of a preexisting medical condition (other than the condition that is being treated by the trial) following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. The number of participants experiencing such adverse events that are related to the study drug are reported here.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 20
Participants | 15

3. Secondary Outcome: Number of Participants With Overall Response
Description: Response was evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Overall response is defined as the proportion of participants whose disease either decreased (partial response- PR) or disappeared (Complete response - CR).
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=20)
Infection - Other (Infections and infestations) | 1 (1) — Hospital acquired nosocomial S. aureus infection
Dehydration (Gastrointestinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Pain (Nervous system disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1) — Urinary Tract Infection
Renal Failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=20)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Fatigue (General disorders) | 7 (7)
Nausea/Vomiting (Gastrointestinal disorders) | 3 (3)
Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.